CLINICAL TRIAL: NCT04005222
Title: Determine the Effects of Selenium and Melatonin on Ocular Ischemic Syndrome
Brief Title: Effects of Selenium and Melatonin on Ocular Ischemic Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beytepe Murat Erdi Eker State Hospital (Other)
Responsible Party: Principal Investigator, Hande Telek, Ophthalmology, MD,Principal Investigator, Beytepe Murat Erdi Eker State Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BeytepeMuratErdiEkerSH
Record Dates: First submitted 2019-06-24; First posted 2019-07-02 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Anterior Segment Ischemia (Diagnosis)
Keywords: Ocular ischemic syndrome; selenium; melatonin; MDA; GSH
MeSH Terms: conditions — Disease | interventions — Selenium; Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELENIUM (Other): The patients in this group were supplemented with oral selenium at 0.1mg/kg doses twice daily for one month. After selenium supplementation period was completed, AC sampling as described above.
  Interventions: Drug: SELENIUM
- MELATONIN (Other): The patients in this group were supplemented with oral melatonin 0.5 mg/kg/day doses twice daily for one month. After supplementation was completed 0.1 cc sampling from AC.
  Interventions: Drug: MELATONIN

INTERVENTIONS:
Drug: SELENIUM — Increased lipid peroxidation associated with ischemia of the anterior segment has been prevented by selenium supplementation.
  Other Names: MELATONIN
  Arms: SELENIUM
Drug: MELATONIN — Increased lipid peroxidation associated with ischemia of the anterior segment has been prevented by melatonin supplementation.
  Other Names: SELENIUM
  Arms: MELATONIN

SUMMARY:
ABSTRACT:

PURPOSE: To determine the effects of selenium, melatonin and selenium + melatonin administered for one month on anterior chamber (AC ) malondialdehyde (MDA) and AC glutathione (GSH) levels in patients with Ocular ischemic syndrome.

MATERIAL AND METHODS: Thirtyfive patients were included in the study. Study groups were formed as follows: 1-Control group, 2-Ischemia group 3-Selenium Ischemia group, 4-Melatonin Ischemia group, 5-Selenium + Melatonin + Ischemia group. AC samples were obtained. MDA and GSH levels in AC samples were evaluated.

RESULTS : MDA levels were significantly increased in ischemia groups. Selenium and melatonin supplementation resulted in reduction of MDA levels and significant increase in GSH values.

DISCUSSION: Increased lipid peroxidation associated with ischemia of the anterior segment has been prevented by selenium and melatonin supplementation.

KEYWORDS: Ocular ischemic syndrome, selenium, melatonin, MDA, GSH

DETAILED DESCRIPTION:
In this retroprospective study, patients who presented with the clinical features of OIS or who had a history of OIS and who had visited the Department of Ophthalmology or who were referred by the Department of Cardiology were considered for inclusion. The patients of OIS were included according to the following criteria (26-29) (1) when the stenosis of the ipsilateral (to the affected eye) internal carotid artery (ICA) was >50% and the ICA blood flow velocity was abnormal; (2) abnormal ocular symptoms and/or signs that could not be explained by other ocular diseases. The ocular symptoms included amaurosis fugax , visual loss ,floaters, metamorphopsia, phosphenes ,diplopia ,and ocular/periorbital pain . Most patients (88.10%) complained of constitutional symptoms, such as headache, syncope, palpitations, hemiplegia, and claudication.The patients who were suffered from other ocular diseases, including primary glaucoma, uveitis, age-related macular degeneration, symmetrical proliferative diabetic retinopathy, choroidal detachment, retinal detachment, hereditary eye diseases, ocular tumor, or ocular trauma, were excluded. Informed consent was acquired from all of the participants before the collection of clinical materials. The study adhered to the tenets of the Declaration of Helsinki.

All of the OIS patients underwent carotid artery color Doppler imaging (CDI) and/or computed tomographic angiography (CTA) to identify the ICA stenosis. Detailed ophthalmic examinations, including best-corrected visual acuity (BCVA), intraocular pressure (IOP), slit-lamp exam, and funduscopy were performed at each follow-up visit. Constitutional and ocular symptoms, medical history (arterial hypertension, diabetes mellitus (DM), hyperlipidemia (HLP), coronary heart disease, cerebrovascular disease, and so on), the clinical department of the first visit, and treatments were also recorded. A statistical description was generated using SPSS for Windows, version 22.0.

Twenty eight OIS patients were recruited in our study, including 20 males (%71,4) and 8 females (%28,6). The age of onset ranged from 58 to 87 years (65.10 ± 10.95), with the majority of patients aged between 61 and 75 years (69.50%). No statistically significant difference was found for gender and age between groups (p <0,01) The study was conducted at Trabzon Numune Training and Research Hospital between May 2014 and September 2016. Approval from the Trabzon Numune Training and Research Hospital Ethics Committee was obtained. All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

Patients were divided into five groups.

1. Control group: Seven healty person were included in this group. After topical anesthesia approximately 0.1 cc samples were obtained from the anterior chamber.
2. Ischemia group: Seven OIS patients were included in this group. Under topical anesthesia, 0.1 cc samples were obtained from the AC.
3. Selenium + Ischemia group: Seven OIS patients were included in this group. The patients in this group were supplemented with oral selenium at 0.1mg/kg doses twice daily for one month. After selenium supplementation period was completed, AC sampling as described above.
4. Melatonin + Ischemia group: Seven OIS patients were included in this group. The patients in this group were supplemented with oral melatonin 0.5 mg/kg/day doses twice daily for one month. After supplementation was completed 0.1 cc sampling from AC.
5. Selenium + Melatonin + Ischemia group: Seven OIS patients were included in this group . The patients were supplemented with selenium and melatonin for one month as described above, subsequently 0.1 cc sampling from AC.

In order to determine AC Malondialdehyde (MDA) levels, 2.5 ml of 10% TCA (tricholoroessigaurekrist.) was put in a test tube, 0.1 ml of AC sample from the patients was added. Tubes were vortexed and sealed. Incubation was applied for 15 minutes in 90ºC water bath. They were cooled in cold water and their absorbance values were read with reference to blank on spectrophotometer at 532 nm. Results were presented as nmol/ml. At the beginning of the testing, blank was prepared by placing the same amount of distilled water instead of plasma in the blank tube and performing the same procedures. In order to measure AC Glutathione (GSH) levels, AC samples placed in tubes containing EDTA were centrifuged at 3000 rpm for 5 minutes. The samples were washed 3 times with 0.9% saline solution and 50μl of each sample was derived. Consecutively, 450μl of distilled water and 500μl of 10% sulfosalicylic acid were added. The mixture was cooled in ice for 1 hour and then centrifuged at 4000 rev for 3 minutes. Subsequently, 200μl of the supernatant was derived and consecutively 8 ml of phosphate buffer with pH of 6.8, 78 μl of 1 N NaOH and 100μl of Ellman solution were added. After waiting for 5 minutes, absorbance values in reagent tube were read with reference to distilled water on spectrophotometer at 412 nm.Ellman solution was prepared by dissolving 100 mg of 5'-5'-dithiobis-2-nitrobenzoic acit (DTNB) in 100 ml of pH 7.8 phosphate buffer. Glutathione standard was prepared as 15.34mg/100 ml by dissolving 15.34 mg of reduced glutathione in 100 ml of 1 nm sodium EDTA. Results were presented as mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* The patients of Ocular ischemic syndrome (OIS) were the stenosis of the ipsilateral (to the affected eye) internal carotid artery (ICA) was >50%
* The patients of Ocular ischemic syndrome (OIS) who the ICA blood flow velocity was abnormal;
* Abnormal ocular symptoms and/or signs that could not be explained by other ocular diseases.

Exclusion Criteria:

* The patients who were suffered from other ocular diseases( primary glaucoma, uveitis, age-related macular degeneration, symmetrical proliferative diabetic retinopathy, choroidal detachment, retinal detachment, hereditary eye diseases, ocular tumor, or ocular trauma)

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To determine the effects of selenium on anterior chamber (AC ) malondialdehyde (MDA) and AC glutathione (GSH) levels in patients with Ocular ischemic syndrome | The patients were supplemented with oral selenium for one month.
  The patients were supplemented with oral selenium at 0.1mg/kg doses twice daily for one month. After selenium supplementation period was completed, 0.1 cc samples were obtained from the anterior chamber (AC). And then determine AC Malondialdehyde (MDA) and Glutathione (GSH) levels.
To determine the effects of melatonin on anterior chamber (AC ) malondialdehyde (MDA) and AC glutathione (GSH) levels in patients with Ocular ischemic syndrome | The patients were supplemented with oral melatonin for one month.
  The patients in this group were supplemented with oral melatonin 0.5 mg/kg/day doses twice daily for one month. After supplementation was completed 0.1 cc sampling from AC. And then determine AC Malondialdehyde (MDA) and Glutathione (GSH) levels.

REFERENCES:
- [Derived] Telek HH. Effects of Selenium and Melatonin on Ocular Ischemic Syndrome. Biomed Res Int. 2019 Dec 6;2019:8080564. doi: 10.1155/2019/8080564. eCollection 2019. PMID 31886253